CLINICAL TRIAL: NCT02253849
Title: A Single Centre, Open-label Study With Healthy Adult Volunteers to Determine the Effects of Single-dose and Steady-state TPV/r 500/200 mg on the Steady-state Pharmacokinetics of Carbamazepine (200 mg Twice Daily)
Brief Title: Effects of TPV/r on the Pharmacokinetics of Carbamazepine in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1182.80
Record Dates: First submitted 2014-09-30; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — Carbamazepine; tipranavir; Ritonavir

ARMS (1):
- CBZ - TPB/r+CBZ (Experimental): Days 1-14: carbamazepine (CBZ) twice daily
  Days 15-22: CBZ twice daily plus TPV/r twice daily
  Interventions: Drug: Carbamazepine; Drug: Tipranavir; Drug: Ritonavir

INTERVENTIONS:
Drug: Carbamazepine
Drug: Tipranavir
Drug: Ritonavir

SUMMARY:
Study to assess the steady-state pharmacokinetics of carbamazepine (CBZ) at 200 mg or 100 mg twice daily, depending on tolerability, and administered alone and in combination with tipranavir/ritonavir (TPV/r) after a single dose (500/200 mg) and at steady-state (500/200 mg twice-daily)

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and non-pregnant, non-lactating female subjects as determined by results of screening
* Signed written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* The ability to understand and sign a written informed consent form, prior to participation in any screening procedures and must be willing to comply with all study requirements
* Age >19 and <59 years
* Weight ≥ 60 kg
* BMI >18.5 and <35 kg/m2
* Ability to maintain adequate contraception if applicable

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate, and electrocardiogram) deviating from normal and of clinical relevance
* AV block including 1°
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, haematological, oncological or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Relevant history of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Known hypersensitivity to TPV, Ritonavir (RTV), carbamazepine or antiretroviral drugs (marketed or experimental use as part of clinical research studies)
* Known elevated liver enzymes in past trials with any compound
* Intake of drugs with a long half-life (>24 hours) (<1 month prior to administration or during the trial)
* Prescription or over the counter medications (including vitamins, minerals, herbal supplements and antacids), dietary supplements 14 days prior to study drug administration or expected during the trial)
* Participation in another trial with an investigational drug (<2 months prior to administration or expected during trial)
* Smoker with a consumption of >10 cigarettes or >3 cigars or >3 pipes/day and those who cannot keep tobacco intake constant
* Alcohol abuse (>60 g/day)
* Drug abuse
* Blood donation or loss >400 mL, <1 month prior to administration or expected during the trial
* Clinically relevant laboratory abnormalities
* Inability to comply with dietary regimen of study centre

For female subjects:

* Pregnancy or planning to become pregnant within 60 days of study completion
* Positive pregnancy test
* Have not been using a barrier method of contraception for at least 3 months prior to participation in the study
* Are not willing or are unable to use a reliable method of barrier contraception (such as diaphragm with spermicidal cream/jelly or condoms with spermicidal foam), during and up to 2 months after completion/termination of the trial
* Chronic use of oral contraception or hormone replacement containing ethinyl estradiol
* Breast-feeding

Ages: 20 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2005-11; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of Carbamazepine in plasma over the time interval t0h to t12h (AUC0-12h) | up to 12 hours after drug administration
Maximum measured concentration of Carbamazepine in plasma (Cmax) | up to 12 hours after drug administration
Drug concentration of Carbamazepine in plasma at 12 hours after drug administration (Cp12h) | up to 12 hours after drug administration

SECONDARY OUTCOMES:
AUC0-12h | up to 12 hours after drug administration
Cmax | up to 12 hours
Cp12h | up to 12 hours after drug administration
Clearance (CL/F) | up to 12 hours after drug administration
Volume of distribution | up to 12 hours after drug administration
Time from dosing to the maximum concentration (Tmax) | up to 12 hours after drug administration
t1/2 (terminal elimination half-life) | up to 12 hours after drug administration
Number of subjects with adverse events | up to 35 days
Number of subjects with clinically relevant changes in laboratory parameters | up to 35 days